CLINICAL TRIAL: NCT06798415
Title: The Clinical Effect of Intralesional Injection of Metronidazole for the Management of Cutaneous Leishmaniasis: Single-arm Open-label Trial
Brief Title: Intralesional Injection of Metronidazole for the Management of Cutaneous Leishmaniasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hayder Adnan Fawzi (Other)
Responsible Party: Sponsor-Investigator, Hayder Adnan Fawzi, Ass Prof, Al-Mustafa University College
Organization: Al-Mustafa University College (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALM25-003; apporval no (69) (Other: Research Ethical Approval of Mustansiriyah University/ College of Pharmacy)
Record Dates: First submitted 2025-01-17; First posted 2025-01-29 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intralesional metronidazole (Experimental): Intralesional metronidazole (5 mg/ml, 100 ml, Flagyl®, Sanofi, France) will be injected into each lesion based on its size (5 mg/cm2). The infiltration of intralesional dose will be given once weekly for up to 6 weeks. Treatment will be stopped in patients cured before 6 weeks of treatment, and patients will be only asked to come for lesion assessment. A fine insulin needle will be used to infiltrate the lesion.
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Intralesional metronidazole (5 mg/ml, 100 ml, Flagyl®, Sanofi, France) will be injected into each lesion based on its size (5 mg/cm2). The infiltration of intralesional dose will be given once weekly for up to 6 weeks. Treatment will be stopped in patients cured before 6 weeks of treatment, and patients were only asked to come for lesion assessment. A fine insulin needle will be used to infiltrate the lesion.
  The lesion will be thoroughly infiltrated with the drug solution until the base will be completely blanched. Depending on the lesion size, the amount of solution required ranged from 0.2 to 4.0 ml per lesion. No local anesthesia will be added. The solutions will be injected intralesionally and not subcutaneously.

SUMMARY:
Aim of the study to evaluate the effectiveness of intralesional metronidazole 0.5% solution as a local injection in treating cutaneous leishmaniasis.

In an open-label single-arm clinical trial, all patients will be given intralesional levofloxacin injections; the patients had cutaneous leishmaniasis lesions. Each lesion will be considered a case in the final analysis. Each lesion will be followed up for 90 days (censor endpoint) or until the lesions are cured.

Intralesional metronidazole (5 mg/ml, 100 ml, Flagyl®, Sanofi, France) will be injected into each lesion based on its size (5 mg/cm2). The infiltration of intralesional dose will be given once weekly for up to 6 weeks. Treatment will be stopped in patients cured before 6 weeks of treatment, and patients will be only asked to come for lesion assessment. A fine insulin needle will be used to infiltrate the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single or multiple (less than seven lesions) lesions of cutaneous leishmaniasis

Exclusion Criteria:

* Immunocompromised
* Allergic reaction to treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate | From enrollment to the end of treatment up to 90 days.
  Patients were followed weekly up to 90 days after the first injection; four parameters were used for assessment as follows according to Sharquie modified leishmania score: 1. Measure the size of the lesion through the surface area 2. Measurement of the induration of the lesion 3. Assess the degree of erythema of the lesion 4. Assess the presence and absence of ulceration The obtained data is converted from numbers into scores. The total score was calculated by adding individual scores. Score 13-16: Mild response. Score 9-12: Moderate response. Score 5-8: Marked response. Score 0-4: Complete response & clearance Both marked and complete responses are considered as a cure

CONTACTS AND LOCATIONS:
Locations (1):
- Mustansiriyah University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided